CLINICAL TRIAL: NCT02129998
Title: The Role of Luteal Progesterone and Preimplantation Factor (PIF) for Successful Implantation and On-going Pregnancy in Assisted Reproductive Technology
Brief Title: The Role of Progesterone and PIF for Successful Implantation and On-going Pregnancy in Assisted Reproductive Technology
Status: Completed | Type: Observational
Sponsor: Regionshospitalet Viborg, Skive (Other)
Collaborators: Ferring Pharmaceuticals (Industry); BioIncept LLC (Industry)
Responsible Party: Principal Investigator, Peter Humaidan, Professor, DMSc, Regionshospitalet Viborg, Skive
Other Study IDs: Progesterone/PIF_Skive
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Infertility
Keywords: Infertility; IVF/ICSI; Progesterone; Preimplantation Factor (PIF)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Embryo culture media
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard IVF/ICSI treatment
  Interventions: Other: IVF/ICSI treatment

INTERVENTIONS:
Other: IVF/ICSI treatment

SUMMARY:
The aim of this study is to achieve a more profound understanding of the endocrine alteration in luteal progesterone level after gonadotrophin stimulated IVF/ICSI cycles and to explore the optimal progesterone level needed for securing implantation and development of early pregnancy.

The second part of the project will determine the value of Preimplantation Factor (PIF) measurement in embryo culture medium as a possible tool for improved embryo selection and the use of PIF as an early pregnancy serum marker for healthy implantation and embryo development.

IVF: In vitro fertilisation, ICSI: Intracytoplasmic sperm injection.

ELIGIBILITY:
Inclusion Criteria:

-All women undergoing IVF/ICSI treatment at the participating clinics in either antagonist protocol or long agonist protocol will be offered participation.

Exclusion Criteria:

-Prior participation in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing IVF/ICSI treatment at 4 Danish Fertility Centres.
Sampling Method: Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
On-going pregnancy rate | 10th week of gestation

SECONDARY OUTCOMES:
Implantation rate | 7th week of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic Skive, Skive, Denmark

REFERENCES:
- [Derived] Thomsen LH, Kesmodel US, Erb K, Bungum L, Pedersen D, Hauge B, Elbaek HO, Povlsen BB, Andersen CY, Humaidan P. The impact of luteal serum progesterone levels on live birth rates-a prospective study of 602 IVF/ICSI cycles. Hum Reprod. 2018 Aug 1;33(8):1506-1516. doi: 10.1093/humrep/dey226. PMID 29955789